CLINICAL TRIAL: NCT02682225
Title: A Single-Center, Single-Dose, Double-Blind, Double-Dummy, Placebo-Controlled, Randomized Crossover Study to Evaluate the Abuse Potential of Intranasal Esketamine Compared to Racemic Intravenous Ketamine in Nondependent, Recreational Users of Perception-Altering Drugs
Brief Title: Crossover Study to Evaluate the Abuse Potential of Intranasal Esketamine Compared to Racemic Intravenous Ketamine in Nondependent, Recreational Drug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108104; 54135419TRD1015 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-02-10; First posted 2016-02-15 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Drug Abuse
Keywords: Esketamine; Placebo; Racemic ketamine; Pharmacokinetics
MeSH Terms: conditions — Substance-Related Disorders | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1: Qualification Session (Experimental): Participants will receive Treatment A (intravenous placebo and intranasal placebo concurrently) on Day 1 and Treatment B (0.5 milligram per kilogram (mg/kg) of intravenous racemic ketamine and intranasal placebo concurrently) on Day 2.
  Interventions: Drug: Intravenous placebo; Drug: Intranasal placebo; Drug: Intravenous racemic ketamine
- Sequence 2: Qualification Session (Experimental): Participants will receive Treatment B (0.5 mg/kg of intravenous racemic ketamine and intranasal placebo concurrently) on Day 1 and Treatment A (intravenous placebo and intranasal placebo concurrently) on Day 2.
  Interventions: Drug: Intravenous placebo; Drug: Intranasal placebo; Drug: Intravenous racemic ketamine
- Sequence 3: Treatment Phase (Experimental): Participants in Sequence 3 will receive Treatment A (intravenous placebo and intranasal placebo) on Day 1 of period 1, Treatment D (intravenous placebo and intranasal 112 milligram (mg) of esketamine as 4 devices, each with 28 mg esketamine) on Day 1 of period 2, Treatment B (0.5 mg/kg of intravenous racemic ketamine and intranasal placebo) on Day 1 of period 3, Treatment C (intravenous placebo and intranasal 84 mg esketamine as 3 devices, each with 28 mg esketamine followed by 1 device with placebo) on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 7 to 14 days.
  Interventions: Drug: Intravenous placebo; Drug: Intranasal placebo; Drug: Intravenous racemic ketamine; Drug: Esketamine 112 mg; Drug: Esketamine 84 mg
- Sequence 4: Treatment Phase (Experimental): Participants in Sequence 4 will receive Treatment B on Day 1 of period 1, Treatment A on Day 1 of period 2, Treatment C on Day 1 of period 3, Treatment D on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 7 to 14 days.
  Interventions: Drug: Intravenous placebo; Drug: Intranasal placebo; Drug: Intravenous racemic ketamine; Drug: Esketamine 112 mg; Drug: Esketamine 84 mg
- Sequence 5: Treatment Phase (Experimental): Participants in Sequence 5 will receive Treatment C on Day 1 of period 1, Treatment B on Day 1 of period 2, Treatment D on Day 1 of period 3, Treatment A on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 7 to 14 days.
  Interventions: Drug: Intravenous placebo; Drug: Intranasal placebo; Drug: Intravenous racemic ketamine; Drug: Esketamine 112 mg; Drug: Esketamine 84 mg
- Sequence 6: Treatment Phase (Experimental): Participants in Sequence 6 will receive Treatment D on Day 1 of period 1, Treatment C on Day 1 of period 2, Treatment A on Day 1 of period 3, Treatment B on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 7 to 14 days.
  Interventions: Drug: Intravenous placebo; Drug: Intranasal placebo; Drug: Intravenous racemic ketamine; Drug: Esketamine 112 mg; Drug: Esketamine 84 mg

INTERVENTIONS:
Drug: Intravenous placebo — Participants will receive placebo, 40-minute, intravenous infusion on Day 1 of Sequence 1, on Day 2 of Sequence 2, on Day 1 of Period 1 in Sequence 3, 5 and 6, on Day 1 of Period 2 in Sequence 3, 4 and 6, on Day 1 of Period 3 in Sequence 4, 5 and 6, and on Day 1 of Period 4 in Sequence 3, 4 and 5.
Drug: Intranasal placebo — Participants will receive placebo, intranasally, on Day 1 or Day 2 in Sequence 1 and 2, on Day 1 of Period 1 in Sequence 3 and 4, on Day 1 of Period 2 in Sequence 4 and 5, on Day 1 of Period 3 in Sequence 3 and 6 and on Day 1 of Period 4 in Sequence 5 and 6.
Drug: Intravenous racemic ketamine — Participants will receive 0.5 mg/kg racemic ketamine, intranasally, on Day 2 in sequence 1, on Day 1 in sequence 2, on Day 1 of Period 1 in Sequence 4, on Day 1 of Period 2 in Sequence 5, on Day 1 of Period 3 in Sequence 3, and on Day 1 of Period 4 in Sequence 6.
Drug: Esketamine 112 mg — Participants will receive 112 mg of Esketamine, intranasally, on Day 1 of Period 1 in Sequence 6, on Day 1 of Period 2 in Sequence 3, on Day 1 of Period 3 in Sequence 5, and on Day 1 of Period 4 in Sequence 4.
  Arms: Sequence 3: Treatment Phase; Sequence 4: Treatment Phase; Sequence 5: Treatment Phase; Sequence 6: Treatment Phase
Drug: Esketamine 84 mg — Participants will receive 84 mg of Esketamine, intranasally, on Day 1 of Period 1 in Sequence 5, on Day 1 of Period 2 in Sequence 6, on Day 1 of Period 3 in Sequence 4, and on Day 1 of Period 4 in Sequence 3.
  Arms: Sequence 3: Treatment Phase; Sequence 4: Treatment Phase; Sequence 5: Treatment Phase; Sequence 6: Treatment Phase

SUMMARY:
The primary objective of this study is to evaluate the abuse potential of intranasal esketamine (112 milligram and 84 mg) compared to racemic intravenous ketamine (0.5 mg/kg) in nondependent, recreational polydrug users of perception-altering drugs.

DETAILED DESCRIPTION:
This is a single-center, single-dose, double-blind, double-dummy, placebo-controlled (participants are randomly assigned to a test treatment or to an identical-appearing treatment that does not contain the test drug), randomized (study medication assigned to participants by chance), crossover study in up to 120 men and women self-identifying as current, recreational, nondependent polydrug users. The study has a Screening Phase (consisting of a Screening Visit and a Qualification Session) and a Treatment Phase. In the Qualification Session participants will be randomized to receive Sequence 1: intravenous placebo and intranasal placebo concurrently (Treatment A) on Day 1 and an intravenous dose (0.5 mg/kg) of racemic ketamine and intranasal placebo concurrently (Treatment B) on Day 2, or the participants will receive Sequence 2: Treatment B on Day 1 and Treatment A on Day 2. In the Treatment Phase eligible participants will be administered 4 treatments: A, B, C (intravenous placebo and intranasal 84 mg esketamine as 3 devices, each with 28 mg esketamine followed by 1 device with placebo) and D (intravenous placebo and intranasal 112 mg of esketamine as 4 devices, each with 28 mg esketamine) in a cross-over manner (1 treatment per period) in Sequence 3, 4, 5, or 6. Periods 1, 2, 3, and 4 will be separated by 7 to 14 days. Primarily the drug abuse potential will be evaluated. Safety of the participants will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (inclusive), and body weight not less than 50 kg
* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study, including the pharmacogenomic research component of the study
* Be a current, recreational, nondependent, polydrug user defined as nonmedical use with at least 2 types of perception-altering drugs of abuse (example, lysergic acid diethylamide, cannabinoids, ketamine, ecstasy/3,4-methylenedioxy-methamphetamine, phencyclidine, psilocybin, and ring-substituted amphetamines with perception altering effects) and at least 10 total lifetime occasions of use with perception-altering drugs of abuse and who like their effects
* Report having used ketamine at least once in a lifetime without moderate or severe adverse effects
* Report having used a perception-altering drug (example, lysergic acid diethylamide, cannabinoids, ketamine, ecstasy/3,4-methylenedioxy-methamphetamine, phencyclidine, psilocybin, and ring substituted amphetamines with perception altering effects) at least once within 3 months prior to the screening phase without moderate or severe adverse effects

Exclusion Criteria:

* Participant with a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic disease, infection, hypertension or vascular disorder, kidney or urinary tract disturbances, sleep apnea, myasthenia gravis, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant has a current or prior diagnosis of psychotic or bipolar disorder
* Participant with clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center (Day -1 of the Qualification Session and each period of the Treatment Phase) as determined by the investigator
* Participant with a history or presence of drug (excluding nicotine or caffeine) or alcohol dependence according to the 4th edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
* Participation in treatment for substance-related disorders within 3 years prior to Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in abuse potential based on Visual Analog Scale | up to Day 2 Period 4 in Treatment Phase
  The abuse potential will be assessed based on visual analog scale (VAS). The VAS score will include for Balancing Measures, Positive and Negative effect at the moment, Perceptual / Dissociative Effects and others).

SECONDARY OUTCOMES:
Change From Baseline in Clinician-Administered Dissociative States Scale (CADSS) Score | up to Day 2 Period 4 in Treatment Phase
  The CADSS is a clinician administered rating scale designed to measure dissociative symptoms. The CADSS comprises 23 subjective items, divided into 3 components: depersonalization, derealization and amnesia. Participant's responses are coded on a 5-point scale (0 = "Not at all" through to 4 = "Extremely). Higher scores indicate worsening
Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Score | up to Day 2 Period 4 in Treatment Phase
  The C-SSRS is a clinical interview to assess severity and track suicidal events providing a summary of both suicidal ideation and behavior to identify the level and type of suicidality present.
Percentage of Participants with Serious Adverse Events (SAEs) and Adverse Events (AEs) | Screening to follow-up visit (11 to 13 days after last dose of study medication)
Maximum Observed Plasma Concentration (Cmax) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  Cmax is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUClast) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  The AUClast is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration
Area Under the Plasma Concentration-Time Curve From Time Zero to 12 Hours (AUC [0-12]) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  The AUC (0-12) is the area under the plasma concentration-time curve from time 0 to 12 hours post-dose.
Elimination Half-Life Period (T1/2) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  T1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
First-order Rate Constant | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  First-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Total Body Clearance (CLT/F) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  Total body clearance will be calculated as dose/AUC(INF). AUC(INF) will be estimated as AUC(0-T) + Ct/λ z, where λ z is the terminal elimination rate constant and Ct is the last observable concentration
Volume of Distribution (Vd/F) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
  The Vd/F is defined as Dose/[Lambda (z)*AUC (0-infinity)].
Cmax Metabolite to Parent Ratio (MPR Cmax) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
AUC(last) Metabolite to Parent Ratio (MPR AUC[last]) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
AUC (infinity) Metabolite to Parent Ratio (MPR AUC [infinity]) | Predose, 0.17, 0.33, 0.5, 0.67, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours post-dose on Day 1
Change from baseline in Nasal Tolerability Questionnaire | up to Day 2 in Period 4 of Treatment Phase
  Participants need to complete a nasal tolerability questionnaire from Screening to end of the study. The questionnaire will be containing different type symptoms with rating (None, mild, moderate and severe).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208